CLINICAL TRIAL: NCT00635505
Title: Randomized, Placebo-Controlled, Parallel, Multi-Center, 12-Week Study to Evaluate the Efficacy and Safety of Albuterol HFA Versus the Active Control, Proventil(R)-HFA in Adult and Adolescent Asthmatic Patients
Brief Title: Controlled, 12-Week Study of Albuterol HFA Versus the Active Control, Proventil(R)-HFA in Asthmatic Patients
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: IND voluntarily withdrawn, without prejudice
Sponsor: Amphastar Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: API-A004-CLN-C
Record Dates: First submitted 2008-03-07; First posted 2008-03-13 (Estimated); Last update posted 2013-07-15 (Estimated); Status verified 2012-07

CONDITIONS: Asthma
Keywords: Asthma; albuterol; HFA
MeSH Terms: conditions — Asthma | interventions — Albuterol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- T (Experimental): albuterol HFA 180 mcg QID
  Interventions: Drug: albuterol HFA (Armstrong's)
- R (Active Comparator): 180 mcg QID 12 weeks
  Interventions: Drug: albuterol HFA (Proventil HFA)
- P (Placebo Comparator): 2 actuations QID 12 weeks or until use of rescue drug
  Interventions: Drug: HFA placebo

INTERVENTIONS:
Drug: albuterol HFA (Armstrong's) — 180 mcg QID 12 weeks
  Arms: T
Drug: albuterol HFA (Proventil HFA) — 180 mcg QID 12 weeks
  Other Names: Proventil HFA
  Arms: R
Drug: HFA placebo — 2 actuations QID 12 weeks or until use of rescue drug
  Arms: P

SUMMARY:
This 12-week clinical study evaluates the safety and efficacy of Albuterol Sulfate HFA Inhalation Aerosol (Albuterol-HFA, or: A004), Armstrong's proposed HFA formulation of metered dose inhaler (MDI) of Albuterol (Treatment T), in comparison with:

1. Placebo control: (HFA propellant only, Treatment P); and
2. Active control: 3M/Key's Proventil-HFA (Treatment R).

The treatments will be given as self-administered oral inhalations in adult and adolescent patients with mild-to-moderate asthma, for 12-weeks. Dosing regimen throughout the 12-week study is two actuations four times daily (QID).

DETAILED DESCRIPTION:
This is a randomized, parallel, multicenter, 12-week study in adolescent and adult patients with mild-to-moderate asthma, to evaluate the efficacy and safety of Armstrong's Albuterol-HFA MDI, in comparison to a Placebo Control and an Active Control of Proventil-HFA. While Albuterol-HFA (Treatment T) and Placebo (Treatment P) will be double-blinded to both the subjects and investigational staff, the active comparator drug, Proventil-HFA (Treatment R), can only be evaluator-blinded, due to: (1) its physical appearance differing from that of the T and P devices; and (2) unavailability of a Proventil-HFA placebo which would otherwise be used for a double-dummy design. All study medications will have the canisters and all product-identifying text or graphics (e.g., molded text on actuator) masked so that the treatments cannot be identified. No subject in any study arm will be given any information that could reveal the nature of the treatment given. All study subjects will be instructed not to reveal or discuss the study medications to the study staff or other subjects. The designated study evaluator(s), who conduct the clinical visits and safety and efficacy evaluations and perform the data recording and transcription, will be blinded to the study medications.

All subjects will be screened for enrollment, and will be randomized into the following three treatment groups in a double-blinded (for Treatments T and P) or evaluator-blinded (for Treatment R) manner:

Treatment T (Albuterol-HFA, N=200): 216 mcg albuterol sulfate (equivalent to 180 mcg albuterol base), QID; Treatment R (Proventil-HFA, N=50): 216 mcg albuterol sulfate (equivalent to 180 mcg albuterol base), QID; Treatment P (Placebo-HFA, N=50): two actuations of placebo, QID.

Randomization is achieved with blocks of six (6), with four (4) patients receiving Albuterol-HFA for every one (1) patient receiving Proventil-HFA and every one (1) receiving the Placebo-HFA. At each Clinical Visit that takes place every 3 weeks, the double-blinded (T, P) or evaluator-blinded (R) study drugs will be distributed in resealable masking pouches to the subjects of each arm.

An additional aim of the study is to evaluate the effect of weekly cleaning on the Albuterol-HFA MDI device clinical performance throughout the four, 3-week life-of-device treatment cycles, in conformance with the FDA's specific requirements.

Arms:

All subjects will be screened for enrollment, and will be randomized into the following three treatment groups in a double-blinded (for Treatments T and P) or evaluator-blinded (for Treatment R) manner:

Treatment T (Albuterol-HFA, N=200): 216 mcg albuterol sulfate (equivalent to 180 mcg albuterol base), QID; Treatment R (Proventil-HFA, N=50): 216 mcg albuterol sulfate (equivalent to 180 mcg albuterol base), QID; Treatment P (Placebo-HFA, N=50): two actuations of placebo, QID.

ELIGIBILITY:
Inclusion Criteria:

* Male and female asthma patients aged 12 - 75 years, in general good health.
* A documented history of mild to moderate asthma, for at-least 6-months prior to Screening, requiring inhaled B2-adrenergic agonists, with or without orally inhaled corticosteroids, for asthma treatment.
* Satisfying criteria of asthma stability, defined as no asthma-related hospitalization or emergency visits, and no significant changes in asthma therapy, over 4 weeks prior to Screening (with exception for switching from long- to short-acting B2-agonists).
* Can tolerate withholding treatment with inhaled bronchodilators and other allowed medications for the minimum washout periods indicated in Appendix II prior to the Screening Baseline FEV1 testing.
* Having a Screening Baseline FEV1 test that falls within 50-90% of the predicted values.
* Airway Reversibility PFT at screening should demonstrate a greater than 12% increase in FEV1 at 30 minutes of inhaling 2 actuations of Ventolin-HFA (180 mcg albuterol base).
* Demonstrating satisfactory techniques in the use of metered-dose inhaler (MDIs) and a hand held peak flow meter.
* Female patients of child-bearing potential being non-pregnant and non-lactating at Screening and throughout the study, and using an acceptable method of contraception during the study.
* Has properly consented to participate in this study.

Exclusion Criteria:

* Male and female asthma patients aged 12 - 75 years, in general good health.
* A documented history of mild to moderate asthma, for at-least 6-months prior to Screening, requiring inhaled B2-adrenergic agonists, with or without orally inhaled corticosteroids, for asthma treatment.
* Satisfying criteria of asthma stability, defined as no asthma-related hospitalization or emergency visits, and no significant changes in asthma therapy, over 4 weeks prior to Screening (with exception for switching from long- to short-acting B2-agonists).
* Can tolerate withholding treatment with inhaled bronchodilators and other allowed medications for the minimum washout periods indicated in Appendix II prior to the Screening Baseline FEV1 testing.
* Having a Screening Baseline FEV1 test that falls within 50-90% of the predicted values.
* Airway Reversibility PFT at screening should demonstrate a greater than12% increase in FEV1 at 30 minutes of inhaling 2 actuations of Ventolin-HFA (180 mcg albuterol base).
* Demonstrating satisfactory techniques in the use of metered-dose inhaler (MDIs) and a hand held peak flow meter.
* Female patients of child-bearing potential being non-pregnant and non-lactating at Screening and throughout the study, and using an acceptable method of contraception during the study.
* Has properly consented to participate in this study.

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2007-09; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is the bronchodilator effect expressed as the mean area under the curve (AUC) of FEV1 (% change from Same-Day Baseline FEV1) versus time. | Concurent with each visit

SECONDARY OUTCOMES:
The comparative analysis of AUC of FEV1 (% change from the Same-Day Baseline) versus time, for bronchodilator effect (between Albuterol-HFA and Proventil-HFA). | End of Study
AUC of FEV1-time curve (changes of actual volumes from the Same-Day Baseline). | End of Study
Time to onset of bronchodilator effect, determined by linear interpolation as the time point where FEV1 first reaches 12% over Same-Day Baseline. | End of Study
The peak bronchodilator response, defined as the maximum FEV1 (% change from Same-Day Baseline) post-dose. | end of study
The time to peak FEV1 effect, measured as the time point of peak response, as defined (4) above. | End of Study
Duration of bronchodilator effect, defined as the total length of time when FEV1 is maintained 12% above the respective Same-Day Baseline values (time points calculated with linear interpolation). | Concurrent with each visit
Percentage of positive responders including those whose FEV1 exceed the Same-Day Baseline by 12% within 30 minutes post-dose (quick responders), and during the entire 6 hr post-dose (overall responders). | Concurrent with visit
Number of inhalations of the rescue inhalers taken. | Concurrent with each visit
Global assessment of Overall Asthma Control Scores by investigators. | End of Study
Total daytime asthma symptom scores. | End of Study
Nighttime sleep disturbance scores. | End of Study
Morning pre-dose Peak Expiratory Flow Rate (PEF). | Concurrent with each visit
The clinical performances of the Albuterol-HFA MDI at the representative first, middle and last one third of the usable life stage, are compared with each other, and are also compared to those of the active control, Proventil-HFA. | End of Study
The in vitro performance of the Albuterol-HFA MDI will be evaluated. | Concurrent with each visit
Vital signs (SBP/DBP, and heart rate) will be monitored at Clinical Visit 1, 3 and 5, at baseline (within 30 minutes prior to dosing), and 90+/-15 min, and 360+/-30 min, post-dose. | concurrent with study visits as noted
A 12-lead ECG (for HR, QT and QTc intervals) will be recorded at Screening Visit, and at baseline (within 30 min) pre-dose and at 90+/-15 min post-dose (predicted time of peak effect). | Clinical Visits 1 and 5
Data for CBC, blood chemistry panel (8-hr fasted), and urinalysis. | Screening and end-of-study
Study compliance and diaries will be reviewed | at all cliniical visits
Concomitant medications will be reviewed and recorded | each study visit
Adverse events/side effects whether observed by investigators or reported by subjects, will be documented, evaluated, followed up, and treated if deemed necessary. | concurrent with each study visit

CONTACTS AND LOCATIONS:
Locations (42):
- United States (42):
  - Pulmonary Associates of Mobile, PC, Mobile, Alabama
  - Allergy & Asthma Specialists Medical Group, Huntington Beach, California
  - Allergy Asthma & Respiratory Care Medical Center, Long Beach, California
  - Allergy & Asthma Care Center, Long Beach, California
  - Southern California Research, Mission Viejo, California
  - CHOC PSF, AMC, Divison AA and I, Orange, California
  - Clinical Trials of Orange County, Orange, California
  - Peninsula Research Associates, Rolling Hills Estates, California
  - Allergy Associates Medical Group, San Diego, California
  - Allergy & Asthma Associates of Santa Clara Valley Research Centere, San Jose, California
  - Bensch Research Associates, Stockton, California
  - Colorado Allergy and Asthma Centers, Denver, Colorado
  - Colorado Allergy and Asthma Centers, Lakewood, Colorado
  - Rocky Mountain center for Clinical Research, Wheat Ridge, Colorado
  - Waterbury Pulmonary Research, Waterbury, Connecticut
  - Allergy and Asthma Care of Florida, Ocala, Florida
  - Brandon-Valrico Center for Allergy and Astham Research,LLC, Valrico, Florida
  - Atlanta Allergy and Asthma Clinic, Woodstock, Georgia
  - Family Allergy and Asthma Research Institute, Louisville, Kentucky
  - Northeast Medical Research Group, North Dartmouth, Massachusetts
  - Park Nicollet Institute, Minneapolis, Minnesota
  - MEDEX Healthcare Research, Inc., St Louis, Missouri
  - The Clinical Research Center, LLC, St Louis, Missouri
  - Clinical Research Group of Montana, Bozeman, Montana
  - Montant Medical Research, Missoula, Montana
  - Asthma and Allergy Center, PC, Papillion, Nebraska
  - New Horizons Clinical Research, Cincinnati, Ohio
  - Toledo Center for Clinical Research, Sylvania, Ohio
  - Integrated Medical Research, Ashland, Oregon
  - Allergy & Asthma Research Group, Eugene, Oregon
  - Allergy Asthma and Dermatology Research, Lake Oswego, Oregon
  - Clinical Research Institute of Southern Oregon, Medford, Oregon
  - Allergy Associates Research Center, Portland, Oregon
  - Allergy and Clinical Immunology Associates, Pittsburgh, Pennsylvania
  - Pharmaceutical Research & Consulting, Inc., Dallas, Texas
  - Allergy and Asthma Associates of Houston, Houston, Texas
  - Clinical Trials of North Houston, Houston, Texas
  - Kerrville Allergy and Asthma Associates, Kerrville, Texas
  - Biogenics Research Institute, San Antonio, Texas
  - Sylvania Research Associates, San Antonio, Texas
  - Virginia Adult and Pediatric Allergy and Asthma, PC, Richmond, Virginia
  - Asthma, Inc., Seattle, Washington